CLINICAL TRIAL: NCT04415580
Title: Effects of Vestibular Rehabilitation in Patients With Severe Traumatic Brain Injury: a Randomized Controlled Trial
Brief Title: Vestibular Rehabilitation and Severe Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Marco Tramontano, head of rehabilitation Services, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FSLCE/PROG.700
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Severe Traumatic Brain Injury; Gait Disorders, Neurologic
MeSH Terms: conditions — Brain Injuries, Traumatic; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabilitation Group (Experimental)
  Interventions: Other: Vestibular Rehabilitation (VR)
- Conventional rehabilitation Group (Active Comparator)
  Interventions: Other: Conventional Neurorehabilitation

INTERVENTIONS:
Other: Vestibular Rehabilitation (VR) — VR consisted of two types of exercises, i.e., those for gaze stability and those for postural stability
  * Gaze stability exercises The patients will perform the exercises while holding their gaze on a firm target (VORx1) during active horizontal and vertical head movements (one minute for each axis).
  * Postural stability exercises March in Place Each patient will ask to get on a foam cushion of 10 cm in height and then will blindfold. Treadmill Training As preparation for training, all subjects underwent a 1-minute walk on treadmill with open eyes using preferred walking speed. Immediately after preparation, patients will blindfold and will ask to walk on treadmill without support of hands for 4 minutes.
  When patients made the mistake of changing direction, the physiotherapist help them to keep the right position using verbal cues (e.g., you are turning left or right).
  Arms: Vestibular Rehabilitation Group
Other: Conventional Neurorehabilitation — muscles stretching, active and assisted limbs mobilization, four limbs coordination exercises, balance training on instable platform and gait training
  Arms: Conventional rehabilitation Group

SUMMARY:
Severe brain injury (sTBI) is one of the most common causes of long-term disability and is considered the most frequent cause of mortality and serious disability in young adults in industrialized countries. It is defined as an alteration of brain function with loss of consciousness in the acute phase for at least 24 hours (Glasgow Coma Scale (GCS) <8) and it can induce a wide range of deficit, including cognitive-behavioural, motors, psychics, language, vision, coordination and balance impairments. Chronic vestibular symptoms such as dizziness and balance deficits (both static and dynamic postural instability) are present in patients with brain injury. These aspects can cause functions limitation and psychological distress, negatively impacting negatively on subjects' quality of life and social reintegration and are considered unfavourable prognostic factors of the recovery process. The literature supports the use of vestibular rehabilitation techniques in patients with mild and moderate brain injury, however, to date, no studies investigated the effect of vestibular rehabilitation in sTBI patients. The main aim of this randomized controlled trail is to verify the effect of a personalized vestibular training on balance and gait disorders in sTBI patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 and 65 years;
* Glasgow coma scale (GCS) score ≤ 8 (used to objectively describe the severity of impaired consciousness at the time of injury)
* Level of cognitive functioning (LCF) ≥7;
* Ability to understand verbal commands and the informed consent.
* Presence of static and dynamic balance impairments.
* Functional Ambulation Classification (FAC) ≥ 3

Exclusion Criteria:

* Glasgow coma scale (GCS) score >8
* Level of cognitive functioning (LCF) <7
* Inability to understand verbal commands
* Absence of static and dynamic balance impairments.
* Functional Ambulation Classification (FAC) < 3

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index Scoring Form (DGI) | Baseline to 8 weeks after the end training
  Change of Dynamic Gait Index Scoring Form (DGI) from baseline at 4 weeks of training, at 4 weeks after the end of the training and after 8 weeks after the end of the training. DGI values ranging from 0 to 24, where 0 means the worse outcome and 24 the best one.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | Baseline to 8 weeks after the end training
  Change of Berg Balance Scale (BBS) from baseline at 4 weeks of training, at 4 weeks after the end of the training and after 8 weeks after the end of the training. BBS values ranging from 0 to 56, where 0 means the worse outcome and 56 the best one
Community Balance & Mobility Scale (CB&M) | Baseline to 8 weeks after the end training
  Change of Community Balance and Mobility Scale (CB&M) from baseline at 4 weeks of training, at 4 weeks after the end of the training and after 8 weeks after the end of the training. CB&M values ranging from 0 to 96, where 0 means the worse outcome and 96 the best one.
Activities-specific Balance Confidence scale (ABC) | Baseline to 8 weeks after the end training
  Change of Activities-specific Balance Confidence scale (ABC) from baseline at 4 weeks of training, at 4 weeks after the end of the training and after 8 weeks after the end of the training. ABC values ranging from 0% to 100%, where 0% means the worse outcome and 100% the best one.
Community Integration Questionnaire (CIQ) | Baseline to 8 weeks after the end training
  Change of Community Integration Questionnaire (CIQ) from baseline at 4 weeks of training, at 4 weeks after the end of the training and after 8 weeks after the end of the training. CIQ values ranging from 0 to 29, where 0means the worse outcome and 29 the best one.
Dizziness Handicap Inventory (DHI) | Baseline to 8 weeks after the end training
  Dizziness Handicap Inventory (DHI) from baseline at 4 weeks of training, at 4 weeks after the end of the training and after 8 weeks after the end of the training. DHI values ranging from 0 to 100, where 100 means the worse outcome and 0 the best one.
Instrumental Assessment | Baseline to 8 weeks after the end training
  Postural and gait functional assessment performed using inertial motion capture systems (Opal, APDM Inc., Portland, Oregon, USA, portable devices controlling 6 inertial/magnetic measurement units providing 3D orientation and kinematic). The assessments were performed at the baseline, 4 weeks of training, at 4 weeks after the end of the training and after 8 weeks after the end of the training

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Marco Tramontano, Roma, Rm
  - Santa Lucia Foundation I.R.C.C.S., Roma, Rm